CLINICAL TRIAL: NCT04725266
Title: A Family-based Intervention for Drug-abusing Adults in Hong Kong: a Quasi-experimental Trial
Brief Title: A Family-based Intervention for Drug-abusing Adults in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Sheng Kung Hui Welfare Council Limited (Other)
Responsible Party: Principal Investigator, Dr.Yik-Wa Law, Associate Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200018
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Drug Abuse
Keywords: drug abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- family-based intervention plus routine care (Experimental): This group of participants including drug abusers and their families will be receiving family-based intervention which is a well-designed intervention with group sessions and routine care provided by professional social workers in local social service center.
  Interventions: Behavioral: Family-based intervention; Other: routine care
- routine care (Active Comparator): The group of participants will receive routine care which is widely used in social service providers and mainly includes individual counselling service for drug abusers.
  Interventions: Other: routine care

INTERVENTIONS:
Behavioral: Family-based intervention — The intervention aims to motivate drug abusers to stay drug abstinence and improve family functioning with the support of their own families. In the component of engagement, we will use effective and appropriate skills to engage clients, understand their concerns, and provide necessary resources to them. In the component of role identification, we will help drug abusers identify their family roles through providing education on family roles and responsibilities. The component of affection is designed to learn affective responsiveness and enhance their emotional bonds with each other, while in the component of competence, we will enhance their competency to take care of the family. The intervention will be conducted in group sessions with 4-6 families per group. A total of 17 sessions will be delivered with 1.5-2 hour for each session (6 sessions for Engagement, 3 sessions for Role identification, 3 sessions for Affection, and 3 sessions for Competence).
  Arms: family-based intervention plus routine care
Other: routine care — Routine care includes individual-session components of engagement, case assessment, drug education, service referral, family support, and etc.

SUMMARY:
To develop a family-based intervention with components of engagement, family roles, affection, and competence and verify its effectiveness on drug abstinence and family functioning for drug-abusing adults in Hong Kong; To compare the difference between family-based intervention and routine care which mainly consists of individual counselling services for drug abusers.

DETAILED DESCRIPTION:
This is a quasi-experimental trial examining the effects of a proposed family-based intervention for drug abusers on motivating them to stay drug abstinence and improve family functioning, in which 40 drug abusers with focal families (including spouses and/or children) will be recruited for intervention group receiving both family-based intervention and routine care and 40 drug abusers without involving family will be recruited for comparison group receiving routine care. In the in-take, drug-abusing subjects will be given a brief introduction and invited to provide basic background information about themselves and families. After filling the informed consent, participants will be assigned to intervention group or comparison group according to whether their family will join sessions together. After drug abusers and families fill in the online questionnaire at the baseline (T0), the intervention group will receive family-based intervention and routine care in one month, while the comparison group will receive only routine care in one month. Both groups will be assessed at two time points after intervention period (T1 = 1-month after baseline; T2 = 2-month after baseline). As hypothesized, the intervention group will show a greater reduction in the primary outcomes of drug use and greater increase in the secondary outcomes of family functioning than the comparison group. A repeated-measures analysis of covariance will be conducted to assess the effects of family-based intervention.

ELIGIBILITY:
Inclusion criteria for intervention group:

1. Adults aged 18 to 55
2. Have used drugs in the past 90 days
3. At the time of case recruitment, the subject is engaged in an intimate relationship with a spouse/partner, or having a child/children
4. Understand oral and written Chinese

Exclusion criteria for intervention group:

1. Taking other treatments during intervention
2. The spouse or child of DA are not available to participate in the program

Inclusion criteria for comparison group:

1. Adults aged 18 to 55
2. Have used drugs in the past 90 days
3. Understand oral and written Chinese

Exclusion criteria for comparison group:

1. Taking other treatments during intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline measurements of drug abstinenceat at 1- and 2-months | Baseline, 1- and 2-months
  Changes in scores on drug abstinence is assessed by Timeline Followback (TLFB) in which participants will report the specific date and time of using drugs in the past one month.
  A higher score suggests a longer time for drug abstinence.
Changes from baseline measurements of frequency of drug use at 1- and 2-months | Baseline, 1-, and 2-months
  Changes in scores on frequency of drug use is measured by Frequency of Drug Use in Past Three Months by Beats Drug Fund.
  A higher score suggests a higher frequency of drug use.

SECONDARY OUTCOMES:
Changes from baseline measurement of marital affection at 1- and 2-months | Baseline, 1- and 2-months
  Changes in scores on marital affection will be measured by the Chinese version of Dyadic Adjustment Scale (C-DAS) with good psychometric properties.
  A higher score on this scale indicates a higher level of marital affection.
Changes from baseline measurement of family functioning at 1- and 2-months | Baseline, 1- and 2-months
  Changes in score on general family functioning will be assessed by Subscale of general functioning of Chinese version of Family Assessment Device (C-FAD). The participants answer each question with a 4-point Likert scale (1=strongly agree, 4=strongly disagree) and the total scores range from 12 to 48.
  A higher score suggests a higher level of family functioning.
Changes from baseline measurement of family roles at 1- and 2-months | Baseline, 1- and 2-months
  Changes in score on family roles will be measured by Perceived Family Responsibility Scale (PFRS) on a 7-point scale ranging from strongly disagree to strongly agree.
  A higher score of family roles suggests that the participants are more responsibility for their families.
Changes from baseline measurement of parenting competency at 1- and 2-months | Baseline, 1- and 2-months
  Changes in score on parenting competence is assessed by Parenting Sense of Competency Scale (PSOC). Parents rate their level of agreement with each item by scores ranging from 1 (strongly disagree) to 6 (strongly agree).
  A higher score indicates a higher level of perceived parenting self-efficacy.
Changes from baseline measurement of mental health at 1- and 2-months | Baseline, 1- and 2-months
  Changes in score on mental health will be assessed by the Chinese version of the Patient Health Questionnaire-9 (PHQ-9) on whether they had been bothered by some mental problems in the past two weeks with a 4-point Likert scale ranging from 1 (not at all) to 4 (nearly every day).
  A higher score suggests a lower level of mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: Yik Wa Law, Principal Investigator — The University of Hong Kong
Locations (1):
- Neo-Horizon of Hong Kong Sheng Kung Hui Welfare Council Limited, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No